CLINICAL TRIAL: NCT04545385
Title: A 16-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Proof-of-Concept Study to Evaluate the Efficacy and Safety of TEV-48574 in Adults With T2-low/Non-T2 Severe Uncontrolled Asthma
Brief Title: A Study to Test if TEV-48574 is Effective in Relieving Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Met pre-specified criteria for futility at interim analysis
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48574-AS-20031; 2020-001927-15 (EudraCT Number)
Record Dates: First submitted 2020-08-24; First posted 2020-09-11 (Actual); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: T2 low, non-T2 asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEV-48574 (Experimental): Participants will receive the investigational medicinal product (IMP) loading doses on the day of randomization and the subsequent corresponding IMP maintenance doses every 2 weeks for a total of 8 doses (1 loading dose and 7 maintenance doses).
  Interventions: Drug: TEV-48574
- Placebo (Placebo Comparator): Participants will receive placebo matching to TEV-48574 SC every 2 weeks for a total of 8 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-48574 — subcutaneous infusion
  Arms: TEV-48574
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the effect of TEV-48574 compared with placebo on loss of asthma control (LoAC) in adult participants with T2-low and non-T2 severe asthma uncontrolled on inhaled corticosteroids plus long-acting beta-agonists (ICS+LABA).

The secondary efficacy objective is to evaluate the effect of TEV-48574 compared with placebo on a range of clinical measures of asthma control.

The duration of participant participation in the study is planned to be up to approximately 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of asthma for at least 12 months prior to the initial screening visit.
* The participant is able to perform technically acceptable and repeatable spirometry, including with a hand-held spirometer, after training
* The participant has had at least one documented clinical asthma exacerbation in the 18 months prior to (but not within 30 days of) the initial screening visit.
* The participant is a non-smoker for ≥6 months with lifetime history ≤10 pack-years, with no current ecigarette or marijuana use.

NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has any concomitant conditions or treatments that could interfere with study conduct.
* The participant is currently pregnant or lactating or is planning to become pregnant during the study.
* The participant has received any live or attenuated vaccine within 15 days of the initial screening visit.

NOTE- Additional criteria apply, please contact the investigator for more information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (97):
- United States (55):
  - Teva Investigational Site 14884, Birmingham, Alabama
  - Teva Investigational Site 14915, Little Rock, Arkansas
  - Teva Investigational Site 14914, Bakersfield, California
  - Teva Investigational Site 15234, Huntington Beach, California
  - Teva Investigational Site 14896, Los Angeles, California
  - Teva Investigational Site 14918, Los Angeles, California
  - Teva Investigational Site 14913, Los Angeles, California
  - Teva Investigational Site 14910, Rolling Hills Estates, California
  - Teva Investigational Site 14907, San Diego, California
  - Teva Investigational Site 14891, San Jose, California
  - Teva Investigational Site 15231, Stockton, California
  - Teva Investigational Site 14916, Walnut Creek, California
  - Teva Investigational Site 14878, Westminster, California
  - Teva Investigational Site 14895, Colorado Springs, Colorado
  - Teva Investigational Site 14917, Denver, Colorado
  - Teva Investigational Site 15222, Coral Gables, Florida
  - Teva Investigational Site 15223, Cutler Bay, Florida
  - Teva Investigational Site 14911, Hialeah, Florida
  - Teva Investigational Site 15225, Hialeah, Florida
  - Teva Investigational Site 14900, Miami, Florida
  - Teva Investigational Site 14883, Miami, Florida
  - Teva Investigational Site 14908, Panama City, Florida
  - Teva Investigational Site 14894, Tallahassee, Florida
  - Teva Investigational Site 15224, Tampa, Florida
  - Teva Investigational Site 14924, Evansville, Indiana
  - Teva Investigational Site 14897, Kansas City, Kansas
  - Teva Investigational Site 15220, Baltimore, Maryland
  - Teva Investigational Site 14877, North Dartmouth, Massachusetts
  - Teva Investigational Site 14922, St Louis, Missouri
  - Teva Investigational Site 14893, St Louis, Missouri
  - Teva Investigational Site 14904, Missoula, Montana
  - Teva Investigational Site 14912, Bellevue, Nebraska
  - Teva Investigational Site 14903, Lincoln, Nebraska
  - Teva Investigational Site 15227, Skillman, New Jersey
  - Teva Investigational Site 15221, Charlotte, North Carolina
  - Teva Investigational Site 15226, Monroe, North Carolina
  - Teva Investigational Site 14882, Raleigh, North Carolina
  - Teva Investigational Site 14887, Wilmington, North Carolina
  - Teva Investigational Site 14889, Cincinnati, Ohio
  - Teva Investigational Site 14886, Dublin, Ohio
  - Teva Investigational Site 14901, Toledo, Ohio
  - Teva Investigational Site 14888, Edmond, Oklahoma
  - Teva Investigational Site 14880, Oklahoma City, Oklahoma
  - Teva Investigational Site 14923, Philadelphia, Pennsylvania
  - Teva Investigational Site 14890, Charleston, South Carolina
  - Teva Investigational Site 14925, Allen, Texas
  - Teva Investigational Site 15230, Austin, Texas
  - Teva Investigational Site 14909, Dallas, Texas
  - Teva Investigational Site 14902, El Paso, Texas
  - Teva Investigational Site 14919, Fort Worth, Texas
  - Teva Investigational Site 14921, Houston, Texas
  - Teva Investigational Site 14905, McKinney, Texas
  - Teva Investigational Site 14879, San Antonio, Texas
  - Teva Investigational Site 14920, Spokane, Washington
  - Teva Investigational Site 14881, Greenfield, Wisconsin
- Bulgaria (13):
  - Teva Investigational Site 59159, Kozloduy
  - Teva Investigational Site 59166, Montana
  - Teva Investigational Site 59163, Plovdiv
  - Teva Investigational Site 59189, Plovdiv
  - Teva Investigational Site 59190, Plovdiv
  - Teva Investigational Site 59164, Rousse
  - Teva Investigational Site 59168, Sofia
  - Teva Investigational Site 59167, Sofia
  - Teva Investigational Site 59160, Stara Zagora
  - Teva Investigational Site 59161, Stara Zagora
  - Teva Investigational Site 59165, Varna
  - Teva Investigational Site 59162, Veliko Tarnovo
  - Teva Investigational Site 59192, Vratsa
- Czechia (6):
  - Teva Investigational Site 54197, Brandýs nad Labem
  - Teva Investigational Site 54194, Jindřichův Hradec
  - Teva Investigational Site 54193, Miroslav
  - Teva Investigational Site 54195, Prague
  - Teva Investigational Site 54203, Strakonice
  - Teva Investigational Site 54196, Teplice
- Germany (12):
  - Teva Investigational Site 32747, Berlin
  - Teva Investigational Site 32759, Frankfurt am Main
  - Teva Investigational Site 32741, Frankfurt am Main
  - Teva Investigational Site 32744, Geesthacht
  - Teva Investigational Site 32739, Hamburg
  - Teva Investigational Site 32746, Hanover
  - Teva Investigational Site 32757, Leipzig
  - Teva Investigational Site 32758, Leipzig
  - Teva Investigational Site 32756, Leipzig
  - Teva Investigational Site 32742, Lübeck
  - Teva Investigational Site 32743, München
  - Teva Investigational Site 32745, Rheine
- Poland (11):
  - Teva Investigational Site 53461, Bydgoszcz
  - Teva Investigational Site 53458, Krakaw
  - Teva Investigational Site 53457, Krakow
  - Teva Investigational Site 53455, Lodz
  - Teva Investigational Site 53483, Poznan
  - Teva Investigational Site 53459, Poznan
  - Teva Investigational Site 53486, Sucha Beskidzka
  - Teva Investigational Site 53462, Tarnów
  - Teva Investigational Site 53485, Warsaw
  - Teva Investigational Site 53460, Wroclaw
  - Teva Investigational Site 53456, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 65 participants were randomly assigned to treatment (33 participants in the TEV-48574 group and 32 participants in the placebo group). Of these, 64 participants received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo matched to TEV-48574 subcutaneously (SC) every 2 weeks for a total of 8 doses.
- TEV-48574: Participants received TEV-48574 loading dose SC on the day of randomization and the subsequent corresponding TEV-48574 maintenance doses SC every 2 weeks for a total of 8 doses (1 loading dose and 7 maintenance doses).
Period: Overall Study
Arm/Group | Placebo | TEV-48574
Started | 32 | 33
Received at Least 1 Dose of Study Drug | 31 | 33
Completed | 17 | 20
Not Completed | 15 | 13
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Loss of asthma control (LoAC) | 0 | 1
Not completed — Study termination | 10 | 10
Not completed — Sponsor decision | 2 | 2
Not completed — Other than specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Placebo: Participants received placebo matched to TEV-48574 SC every 2 weeks for a total of 8 doses.
- Total: Total of all reporting groups
Arm/Group | Placebo | TEV-48574 | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (14.14) | 58.8 (12.38) | 57.6 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 28 | 26 | 54
  Race: Black or African American | 4 | 6 | 10
  Race: Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Loss of Asthma Control (LoAC) During the Treatment Period
Description: The LoAC was defined as any 1 of the following during the treatment period: - morning peak expiratory flow (PEF) decrease ≥30% from baseline on 2 consecutive days or morning handheld forced expiratory volume in the first second of exhalation (FEV1) decrease ≥20% from baseline on 2 consecutive days; - increase in short-acting beta-agonist (SABA)/quick-relief medication ≥6 puffs over baseline use in 24 hours on 2 consecutive days; increase in inhaled corticosteroids (ICS) dose ≥4 × most recent dose; - systemic corticosteroid use; - asthma emergency room (ER) visit or hospitalization.
Time Frame: From randomization (Week 0) until Week 16
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 32 | 33
Participants | 13 | 17
Statistical Analysis 1: Comparison: Placebo vs TEV-48574; Analysis was performed using logistic regression with fixed effects for treatment, baseline FEV1, weight, age group, and gender; Test type: Other; p = 0.7817, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.545 to 4.071]

2. Secondary Outcome: Time From Randomization to LoAC During the Treatment Period
Description: Time (in days) from randomization to LoAC during the treatment period is the interval from randomization to the occurrence of the LoAC. The LoAC was defined as any 1 of the following during the treatment period: - morning PEF decrease ≥30% from baseline on 2 consecutive days or morning handheld FEV1 decrease ≥20% from baseline on 2 consecutive days; - increase in SABA/quick-relief medication ≥6 puffs over baseline use in 24 hours on 2 consecutive days; increase in ICS dose ≥4 × most recent dose; - systemic corticosteroid use; - asthma ER visit or hospitalization.
Time Frame: From randomization (Week 0) until Week 16
Population: The ITT analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 32 | 33
days | NA [60.0 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% confidence interval (CI) could not be calculated. | 109.0 [45.0 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated.

3. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire 6-Question Version (ACQ-6) Score at Week 16
Description: The ACQ-6 is a 6-item validated asthma assessment tool that has been widely used. Six questions are self-assessments (completed by the participant), 5 questions assessing asthma symptoms: night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and 1 question for short-acting bronchodilator use. Each item on the ACQ-6 has a possible score ranges from 0 to 6, and the total score is the mean of all responses. The total score ranging from 0-6 (0=totally controlled and 6=severely uncontrolled). A higher score indicated poorer asthma control.
Time Frame: Baseline, Week 16
Population: The ITT analysis set included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 11 | 16
units on a scale | -0.560 (0.4546) | -0.833 (0.7250)

4. Secondary Outcome: Change From Baseline in Percent Predicted Forced Expiratory Volume in the First Second (FEV1) at Week 16
Description: FEV1 (measured by handheld spirometer) is the volume of air that can be forcibly exhaled from the lungs in the first second. The percent predicted FEV1 equals the participant's observed FEV1 divided by the participant's predicted FEV1 (determined by height and race) and converted to a percentage by multiplying by 100%.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: %predicted FEV1
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 11 | 16
%predicted FEV1 | 0.121 (8.3126) | 4.844 (12.4343)

5. Secondary Outcome: Change From Baseline in Daily Average Use of Short-acting Beta-agonist (SABA) Quick Relief Medication at Week 16
Description: Number of inhalations/puffs of SABA/quick relief inhaler used was recorded in the e-diary daily.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: puffs of SABA/day
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 11 | 16
puffs of SABA/day | -0.235 (1.2641) | -0.305 (1.6501)

6. Secondary Outcome: Number of Participants Who Had a Clinical Asthma Exacerbation (CAE) During the Treatment Period
Description: The CAEs during the study were defined as a worsening of asthma symptoms resulting in any 1 of the following: - the use of systemic corticosteroids (oral or injectable); - an emergency department visit due to asthma treated with systemic corticosteroids; - an inpatient hospitalization due to asthma.
  Worsening asthma included new or increased symptoms or signs that either worried the participant or were related to an asthma-specific alert (if available through the e-diary/handheld spirometer).
Time Frame: From randomization (Week 0) until Week 16
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 32 | 33
Participants | 2 | 3

7. Secondary Outcome: Time From Randomization to First CAE During the Treatment Period for Participants With CAE
Description: as for outcome 6
Time Frame: From randomization (Week 0) until Week 16
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 2 | 3
days | 46.5 [38 to 55] | 37.0 [30 to 54]

8. Secondary Outcome: Change From Baseline in Number of Nighttime Awakenings Due to Asthma at Week 16
Description: Participants recorded the number of nighttime awakenings due to asthma in the e-diary daily, in the morning.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nighttime awakenings
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 11 | 16
nighttime awakenings | -1.224 (2.0182) | -0.208 (2.7274)

9. Secondary Outcome: Percent Change in ICS Dose During the Treatment Period
Description: The ICS dose was not collected in the participant diary as planned.
Time Frame: From randomization (Week 0) until Week 16
Population: Due to change in planned analysis, no data was collected to evaluate this outcome measure.
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Week 16
Description: FVC (measured by handheld spirometer) is the volume of air that can be forcibly and completely blown out after full inspiration, measured in liters.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 11 | 16
liters | 0.014 (0.3052) | 0.155 (0.3964)

11. Secondary Outcome: Change From Baseline in Forced Expiratory Flow at 25-75% of Pulmonary Volume (FEF25%-75%) at Week 16
Description: The FEF25%-75% (measured by handheld spirometer) is the forced expiratory flow from 25% to 75% of FVC
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 11 | 16
liters/second | -0.026 (0.2451) | 0.166 (0.4342)

12. Secondary Outcome: Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) at Week 16
Description: FeNO was performed prior to the on-site spirometry.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 11 | 16
parts per billion (ppb) | 5.364 (6.9609) | 10.375 (12.5850)

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Serious adverse events (SAEs) included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. AEs were considered treatment emergent (TEAEs) if onset occurred on or after the first dose date. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'. AEs include clinically significant changes from baseline in any one of the following categories: clinical laboratory test results, vital signs, ECG findings.
Time Frame: From randomization (Week 0) until Week 24
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-48574
Number analyzed (Participants) | 31 | 33
Participants | 14 | 18

ADVERSE EVENTS:
Time Frame: From randomization (Week 0) until Week 24
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | TEV-48574
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/33
Other Adverse Events (participants affected / at risk) | 4/31 | 6/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | TEV-48574 (N=33)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | TEV-48574 (N=33)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT04545385/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT04545385/SAP_001.pdf